CLINICAL TRIAL: NCT01211509
Title: A Randomized, Double Blind, Placebo Controlled Trial With Montelukast to Treat Bronchiolitis Obliterans Syndrome After Lung Transplantation
Brief Title: Montelukast in Bronchiolitis Obliterans Syndrome
Acronym: MLK002
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Geert Verleden, Prof, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLK002
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Bronchiolitis Obliterans; Lung Transplantation; Graft Rejection
Keywords: montelukast; cysteinyl leukotriene; lung transplantation; bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- montelukast sodium (Experimental): Daily treatment with 10 mg montelukast after diagnosis of fibroproliferative BOS (fBOS) which is the low neutrophilic phenotype within BOS
  Interventions: Drug: Montelukast
- placebo (Placebo Comparator): Lactose monohydricum Ph.Eur.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — After diagnosis of fBOS every day an oral capsule with 10 mg montelukast of placebo
  Other Names: Montelukast TEVA

SUMMARY:
Chronic rejection (or Bronchiolitis Obliterans syndrome-BOS) is a major cause of mortality and morbidity after lung transplantation. Because montelukast has been shown to be of some efficacy in a similar disease (Obliterative Bronchiolitis after bone marrow transplantation), the investigators would like to test if montelukast can indeed slow down the progression of chronic rejection after lung transplantation.

DETAILED DESCRIPTION:
* Prospective, interventional, randomized, double-blind, placebo-controlled trial.
* Clinical setting (tertiary University Hospital).
* Investigator-driven, no pharmaceutical sponsor.
* Lung transplant recipients.
* Add-on of study-drug (placebo or montelukast) to 'standard of care'
* 1:1 inclusion ratio (placebo:montelukast).
* Randomisation at diagnosis of chronic rejection after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fBOS
* Signed informed consent
* Age at least 18 years old at moment of transplantation
* Able to take oral medication

Exclusion Criteria:

* Retransplantation
* Previous organ transplantation
* Multi organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
survival/retransplantation rate after diagnosis of BOS | 1 year after diagnosis
survival/retransplantation rate at 2 years after diagnosis | 2 years after diagnosis

SECONDARY OUTCOMES:
Obstructive and restrictive pulmonary function evolution | during 1 and 2 years of treatment
Bronchoalveolar lavage fluid (BAL) | during 1 and 2 years of treatment
  BAL will be used to assess cellularity, protein and mRNA concentration and microbiology
peripheral blood | during 1 and 2 years of treatment
  peripheral blood will be used to assess C-reactive protein, protein and mRNA concentration and fibrocytes content
Cytomegalovirus (CMV) and non-CMV infection rates | during 1 and 2 years of follow up
Acute rejection and lymphocytic bronchiolitis rates | after 1 and 2 years of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Geert M Verleden, MD, PhD, Principal Investigator — UZ gasthuisberg
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Or R, Gesundheit B, Resnick I, Bitan M, Avraham A, Avgil M, Sacks Z, Shapira MY. Sparing effect by montelukast treatment for chronic graft versus host disease: a pilot study. Transplantation. 2007 Mar 15;83(5):577-81. doi: 10.1097/01.tp.0000255575.03795.df. PMID 17353777
- [Background] Vanaudenaerde BM, Meyts I, Vos R, Geudens N, De Wever W, Verbeken EK, Van Raemdonck DE, Dupont LJ, Verleden GM. A dichotomy in bronchiolitis obliterans syndrome after lung transplantation revealed by azithromycin therapy. Eur Respir J. 2008 Oct;32(4):832-43. doi: 10.1183/09031936.00134307. PMID 18827151